CLINICAL TRIAL: NCT05801120
Title: Effects of Pre-dive Ketone Food Products on Latency to Central Nervous System Oxygen Toxicity
Brief Title: Effects of Pre-dive Ketone Food Products on Latency to CNS Oxygen Toxicity (Aim 1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Navy (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Pro00111000
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Oxygen Toxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketogenic food products one time (Experimental): Dietary Supplement: Ketogenic food products Participants will be given a ketogenic food product prior to the hyperbaric oxygen exposure.
  Interventions: Dietary Supplement: Ketogenic food products
- Experimental: Ketogenic food products two times (Experimental): Dietary Supplement: Ketogenic food products Participants will be given a ketogenic food product prior to the hyperbaric oxygen exposure.
  Interventions: Dietary Supplement: Ketogenic food products
- Experimental: Ketogenic food products three times (Experimental): Dietary Supplement: Ketogenic food products Participants will be given a ketogenic food product prior to the hyperbaric oxygen exposure.
  Interventions: Dietary Supplement: Ketogenic food products

INTERVENTIONS:
Dietary Supplement: Ketogenic food products — Participants will be given a ketogenic food product prior to the hyperbaric oxygen exposure.

SUMMARY:
The purpose of this study is to understand how ketogenic food products affect oxygen toxicity in undersea divers. Oxygen toxicity affecting the central nervous system, mainly the brain, is a result of breathing higher than normal oxygen levels at elevated pressures as can be seen in SCUBA diving or inside a hyperbaric (pressure) chamber. This is a condition that may cause a wide variety of symptoms such as: vision disturbances, ear-ringing, nausea, twitching, irritability, dizziness, and potentially loss of consciousness or seizure. Because nutritional ketosis has been used to reduce or eliminate seizures in humans, it may be beneficial to reduce oxygen toxicity as well. The investigators hope this study will provide a help to develop practical and useful methods for improving the safety of undersea Navy divers, warfighters and submariners.

DETAILED DESCRIPTION:
Central nervous system (CNS) oxygen toxicity continues to be a risk for military divers and constrains their operations. Manifestations of this condition range from nausea, twitching, and tinnitus to seizures and unresponsiveness, and the latter may lead to death by drowning. The NAVY has a need for better methods to prevent or delay the onset of CNS oxygen toxicity (CNSOT) and to safely expand the scope of diving operations. It is the broad objective of this study to generate information that will enhance warfighter safety and performance in relevant NAVY operations by reducing the risk of CNS oxygen toxicity.

It is known that nutritional ketosis through a diet with a high fat-to-carbohydrate ratio (ketogenic diet) can reduce the frequency and severity of epileptic seizures in humans, and a recent animal study has shown that dietary ketosis also delays the onset of CNSOT. In recent years, ketone ester food products ketone esters have been made commercially available which may elevate circulating ketone levels. The investigators aim to investigate whether ketosis from commercially available ketogenic food products prior to a dive will delay the onset of CNSOT.

The first aim of this study will be to determine the effect of ketone food product ingestion on serum ketone levels, and document any relevant side effects. Post-ingestion ketone levels will be trended for 3 different ketone food product regimens in 15 total subjects. Data will be used to select the optimal ketone food product strategy to investigate in the second aim which will be registered separately.

ELIGIBILITY:
Inclusion Criteria:

* Males & females between 18 and 39 years old.
* Predicted (Phase 1) VO2max ≥ 30 ml/kg/min (female) or 35 ml/kg/min (male).
* BMI ≤ 30.0 unless VO2max and baseline exercise profile is deemed appropriate for the study by the PI.

Exclusion Criteria:

* Prolonged QTc on initial ECG
* Currently pregnant or attempting to become pregnant.
* Have a medical history of:

  1. Smoking history deemed significant by PI
  2. Known significant electrolyte disorders
  3. Coronary artery disease
  4. Cardiac arrhythmia deemed significant by PI
  5. Lung disease
  6. Hypertension
  7. Seizures
  8. Exercise intolerance or inability to meet inclusion requirements
  9. Psychiatric disorder deemed significant by PI
  10. Previous pneumothorax or pneumomediastinum
  11. Hypo- or hyperglycemia
  12. Diabetes
  13. Inability to equalize middle ear spaces during hyperbaric compression
  14. Claustrophobia
* Regularly take any medications which may alter heart rate, blood pressure, neurotransmitter function, alter seizure threshold, mood or affect per PI discretion.
* Any other condition limiting ability to perform exercise testing or dive profile as determined by the investigators.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Change in serum acetoacetate levels. | over 6 hours
  Assess serum ketone levels over the course of 6 hours after the ingestion of ketone food products.
Change in beta hydroxybutyrate levels | over 6 hours
Change in acetone levels | over 6 hours

SECONDARY OUTCOMES:
Tolerability of ketone food product ingestion measured by adverse events | 24 hours
  Assessment of side effects which may impair a working diver over a period of 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Derrick, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT05801120/ICF_000.pdf